CLINICAL TRIAL: NCT05369702
Title: Association of Coronary Artery Disease With Lewis and ABO Blood Group Phenotypes- A Case Control Study
Brief Title: Association of Coronary Artery Disease With Lewis and ABO Blood Group Phenotypes
Status: Completed | Type: Observational
Sponsor: Jubilee Mission Medical College and Research Institute (Other)
Responsible Party: Principal Investigator, Sree Raj V, Principal Investigator, Jubilee Mission Medical College and Research Institute
Other Study IDs: 47/19/IEC/JMMC&RI
Record Dates: First submitted 2022-04-29; First posted 2022-05-11 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Coronary Artery Disease
Keywords: ABO blood group system; Lewis negative phenotype; coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CASE(coronary artery disease): Patients with confirmed coronary artery disease
- CONTROL: People without coronary artery disease

SUMMARY:
Primary objective- To study the association of Lewis antigen and A, B, O blood group phenotypes with coronary artery disease patients attending the tertiary care hospital in Kerala.

The secondary objective-To find the association of Lewis antigen and A, B, O blood group phenotypes with smoking, alcohol use, diabetes, hypertension and dyslipidemia.

A case-control study to compare the prevalence of Lewis(a-b-) blood group among confirmed cardiac cases with the prevalence of the same among the general population and thereby find out if individuals with Lewis(a-b-) are more at risk of developing coronary artery disease. This may provide an economical and simple method for identifying subjects at increased risk for coronary artery disease and subsequently lead to more focused preventive measures and eventually to a specific treatment.

ELIGIBILITY:
Inclusion Criteria:

- Patients in the age group of 30-55 years at the time of data collection diagnosed with coronary artery disease based on positive changes in coronary angiogram (more than 70% coronary stenosis)

Exclusion Criteria:

* Patients with other systemic illnesses like malignancy, autoimmune diseases.
* Patients who were not willing to participate in the study.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 70 cases attending the Cardiology department who satisfy the inclusion and exclusion criteria were taken as cases.
  140 (age and gender-matched) healthy blood donors who were eligible to donate blood as per the inclusion and exclusion criteria of Drugs and Cosmetics Rules, 1945 were taken as controls.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of Lewis and ABO blood group phenotypes in cases and controls. | Lewis and ABO phenotype of the study participants was determined immediately after sample collection
  Prevalence Lewis and ABO phenotype in cases will be compared to prevalence of the same in controls.

CONTACTS AND LOCATIONS:
Locations (1):
- Jubilee Mission Medical College & Research Institute, Thrissur, Kerala, India

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-08-14): https://cdn.clinicaltrials.gov/large-docs/02/NCT05369702/Prot_SAP_ICF_000.pdf